CLINICAL TRIAL: NCT07326358
Title: Development and Validation of an Artificial Intelligence System for Anatomic Site Recognition and Lesion Detection Based on Electronic Nasopharyngolaryngoscopic Images: A Prospective Multicenter Study
Brief Title: AI System for Anatomic Recognition & Lesion Detection in Nasopharyngolaryngoscopy: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-811
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Neoplasms; Laryngeal Disease
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Model training and validation cohorts: A deep learning model is trained using the training dataset and validated with the internal validation set.
  Interventions: Other: Diagnostic
- Prospective test cohort: Patients are prospectively enrolled, nasopharyngolaryngoscopy examination videos are collected, and the video data are processed to form a prospective test dataset, which is then used for testing.
  Interventions: Other: Diagnostic

INTERVENTIONS:
Other: Diagnostic — The deep learning model is trained using the training dataset and tested with the internal validation set.
  Groups: Model training and validation cohorts
Other: Diagnostic — The prospective dataset is used for the comparative testing of the model and physicians.
  Groups: Prospective test cohort

SUMMARY:
An artificial intelligence-assisted system is trained and validated by collecting nasopharyngolaryngoscopy images from patients.

DETAILED DESCRIPTION:
To address the clinical pain points of traditional nasopharyngolaryngoscopy, such as incomplete visualization, inaccurate identification, and unclear imaging, this study will retrospectively collect nasopharyngolaryngoscopy images and baseline information (including gender and age) of patients who underwent nasopharyngolaryngoscopy at participating centers for model training and validation. Deep learning algorithms will be applied to construct the model. The final clinical performance evaluation of the model will be conducted using an independent, prospectively collected test cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Underwent standard electronic nasopharyngolaryngoscopy;
* Patients who underwent biopsy sampling have a clear pathological diagnosis;
* Signed a written informed consent form.

Exclusion Criteria:

* Image quality is substandard with severe motion artifacts;
* Lesion images are unclear and incomplete.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Image data of patients who underwent nasopharyngolaryngoscopy and met the research requirements were collected from various sub-centers nationwide.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
performance of lesion detection | Within 3 months after the completion of prospective data collection
  The area under the receiver operating characteristic curve (ROC-AUC) of the model for abnormal lesion detection
performance of anatomic site recognition | Within 3 months after the completion of prospective data collection
  The average precision (AP) of the model for recognizing nasopharyngeal and laryngeal anatomic sites

SECONDARY OUTCOMES:
Comparison of diagnostic performance between the model and physicians | Within 3 months after the completion of prospective data collection
  Differences in sensitivity, specificity, and overall accuracy between the AI model and endoscopists with different years of experience

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided